CLINICAL TRIAL: NCT01342653
Title: Phase II Multicentric Exploratory Single Cohort Clinical Trial to Assess Efficacy and Safety on a New Treatment Scheme by Systemic and Peritoneal Chemotherapy Plus Cytoreduction and HIPEC Plus Adjuvant Treatment in Patients With Peritoneal Carcinomatosis From Gastric Cancer
Brief Title: Clinical Trial at Neoadjuvant Peritoneal and Systemic Chemotherapy Plus HIPEC in Gastric Carcinomatosis
Acronym: HIPEC
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: unable to reach planned recruitment
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-011162-29
Record Dates: First submitted 2011-04-26; First posted 2011-04-27 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Peritoneal Carcinomatosis; Gastric Cancer
Keywords: Peritoneal; Carcinomatosis; Gastric; Cancer; NIPS; HIPEC
MeSH Terms: conditions — Peritoneal Neoplasms; Stomach Neoplasms; Carcinoma; Neoplasms | interventions — Infusions, Parenteral; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NIPS plus HIPEC plus adjuvant chemotherapy (Experimental)
  Interventions: Other: Intraperitoneal and systemic chemotherapy plus maximum cytoreduction plus HIPEC

INTERVENTIONS:
Other: Intraperitoneal and systemic chemotherapy plus maximum cytoreduction plus HIPEC — see Design

SUMMARY:
Implementation of a curative strategy of treatment in peritoneal carcinomatosis of gastric cancer. The goal is to get 1C level of evidence (patient died with "standard" treatment, with this treatment some of them survive) in terms of disease free survival and overall survival.

Methodology: prospective, phase II, multicentric in Spain. Recruitment of 50 patients(to have 31 on treatment) in three years. This strategy is based on neoadjuvant systemic plus simultaneous intraperitoneal and intravenous chemotherapy(NIPS),to treat peritoneal disease by bi-directional approach; next step is cytoreductive surgery and HIPEC. Once patients are discharged, they will follow a systemic adjuvant chemotherapy protocol.

DETAILED DESCRIPTION:
Patients with peritoneal carcinomatosis with gastric cancer who meet all inclusion criteria(and none of exclusion) will follow the next treatment scheme(40 week period of treatment):

Phase I (after one week of peritoneal catheter implant; total treatment 5-8 weeks): intraperitoneal infusion of Docetaxel(30 mg/m2) and Cisplatin (30mg/m2) in 1000 cc of saline. Intravenous administration 5-FU (200 mg/m2/Day, 7 days a week for 2 weeks) simultaneously with 2 cycles of Intraperitoneal administration.

These patients receive between four and six cycles of NIPS. Until phase II 4-6 weeks.

Phase II:cytoreduction (CR) plus HIPEC (total treatment 4 weeks). Maximal efforts to optimum cytoreduction.

HIPEC: intraperitoneal administration: Mytomicin C (15mg/m2)plus Adriamycin (15mg/m2) at 42-43ºC for 60 minutes.

Intravenous simultaneously administration 5-FU (400mg/m2) plus Leucovorin (20mg/m2) for 10 minutes at the beginning of peritoneal perfusion.

Phase III: adjuvant chemotherapy 8-12 weeks after surgery. Those cases reaching optimum cytoreduction (CC0) will be treated with systemic chemotherapy: First day: Docetaxel (75 mg/m2) Cisplatin (75mg/m2). Days 1-5: 5-FU (750mg/m2/d).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-65 years old
* Histological Evidence of peritoneal carcinomatosis from gastric cancer
* No distance metastasis
* ECOG 0-1-2
* No contraindication for complex surgery
* no other malign disease except skin cancer (different from melanoma or cervix cancer CIN III)
* willing to consent and sign ICF.

Exclusion Criteria:

* No Histological Evidence of peritoneal carcinomatosis from gastric cancer
* Previous Gastrectomy due to gastric cancer.
* Patients with gastric cancer and previous systemic chemotherapy
* Peritoneal recurrence due to gastric cancer.
* Distance metastasis
* SP >2 at recruitment or SP>1 at surgery
* previous radiotherapy treatment
* pregnant or breastfeeding women

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 36 months
  patients who reached optimum cytoreduction (CC0)after Phase II and eligible to complete adjuvant treatment(Phase III).

SECONDARY OUTCOMES:
progression free survival | 36 months
overall survival in patients with CC0 | 36 month
overall survival in patients who did not reach optimum cytoreduction | 36 months
morbidity and mortality | first 30 days after surgery procedure
Quality of life after phase I and Phase II | 36 months

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid
  - Centro Oncologico MD Anderson International España, Madrid, Madrid